CLINICAL TRIAL: NCT00411138
Title: Randomized Phase III Trial Comparing Concurrent Chemoradiation and Adjuvant Chemotherapy With Pelvic Radiation Alone in High Risk and Advanced Stage Endometrial Carcinoma: PORTEC-3
Brief Title: Randomized Trial of Radiation Therapy With or Without Chemotherapy for Endometrial Cancer
Acronym: PORTEC-3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University (Other)
Collaborators: Cancer Research UK (Other); Australia New Zealand Gynaecological Oncology Group (Other); NCIC Clinical Trials Group (Network); Mario Negri Institute for Pharmacological Research (Other); UNICANCER (Other)
Responsible Party: Principal Investigator, Carien Creutzberg, Chief Investigator, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000521447; P06.031; CKTO-2006-04 (Other Grant/Funding Number: Dutch Cancer Society); ISRCTN14387080 (Registry Identifier: International Standard Randomised Controlled Trial Number); P06.031-PORTEC-3 (Other: Leiden University Medical Center); 2007-004917-33 (EudraCT Number)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Cancer
Keywords: endometrial clear cell carcinoma; stage II endometrial carcinoma; stage IA grade 3 endometrial carcinoma; stage IB endometrial carcinoma; stage IIIA endometrial carcinoma; stage IIIB endometrial carcinoma; stage IIIC endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy; Brachytherapy; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Therapy (Active Comparator): Pelvic Radiotherapy alone
  Interventions: Radiation: Radiation Therapy
- Radiation Therapy and Chemotherapy (Experimental): Pelvic Radiation plus 2 concurrent cycles cisplatin followed by 4 adjuvant cycles carboplatin and paclitaxel
  Interventions: Radiation: Radiation Therapy; Drug: cisplatin; Drug: carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Radiation Therapy — External beam pelvic radiotherapy (48.6 Gy in 1.8 Gy fractions) Vaginal brachytherapy boost in case of cervical involvement
  Other Names: RT; 3D conformal radiotherapy; IMRT; brachytherapy
Drug: cisplatin — cisplatin 50 mg/m2 i.v., 2 cycles during radiotherapy, 3 wks interval
  Other Names: Cisplatine
  Arms: Radiation Therapy and Chemotherapy
Drug: carboplatin — carboplatin AUC 5, 4 cycles after completion of radiotherapy, 3 wks interval
  Other Names: Carboplatine; Carbotaxol
  Arms: Radiation Therapy and Chemotherapy
Drug: Paclitaxel — paclitaxel 175 mg/m2, 4 cycles after completion of radiotherapy, 3 wks interval
  Other Names: Taxol; Taxolcarbo
  Arms: Radiation Therapy and Chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving chemotherapy together with radiation therapy is more effective than giving radiation therapy alone in treating endometrial cancer.

PURPOSE: This randomized phase III trial is studying chemotherapy and radiation therapy to see how well they work compared with radiation therapy alone in treating patients with high-risk, stage I, stage II, or stage III endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival and failure-free survival of patients with high-risk stage IB-III endometrial carcinoma treated with concurrent chemoradiotherapy followed by adjuvant chemotherapy vs pelvic radiotherapy alone.

Secondary

* Compare the rates of pelvic and distant recurrence, severe (grades 3 and 4) treatment-related toxicity, and quality of life of patients treated with these regimens.

OUTLINE:

This is a multicenter, prospective, open-label, randomized, controlled study. Patients are stratified according to participating group (DGOG vs UK NCRI vs NCIC CTG vs MaNGO vs Unicancer), type of surgery (total abdominal hysterectomy and bilateral salpingo-oophorectomy [TAH-BSO] vs TAH-BSO plus lymphadenectomy vs laparoscopic hysterectomy [TLH-BSO] vs TLH-BSO plus lymphadenectomy), stage (IA vs IB vs II vs III), and histological type (endometrioid carcinoma vs serous or clear cell carcinoma). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive external-beam pelvic radiotherapy 5 days a week for up to 6 weeks, combined with cisplatin IV days 1 and 22. Patients with cervical involvement undergo vaginal brachytherapy boost. At least 3 weeks after completion of chemoradiotherapy, patients undergo adjuvant chemotherapy comprising paclitaxel IV and carboplatin IV on day 1. Adjuvant chemotherapy repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo external-beam pelvic radiotherapy (and vaginal brachytherapy alone in case of cervical involvement) as in arm I.

Quality of life is assessed at baseline, completion of radiotherapy, completion of chemotherapy, at 6 months, and then once a year for 5 years.

After completion of study therapy, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 670 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma, with one of the following postoperative FIGO 2009 stages and grade:

  1. stage IA with invasion, grade 3 with documented LVSI
  2. stage IB grade 3
  3. stage II
  4. stage IIIA or IIIC; or IIIB if parametrial invasion only
  5. stage IA (with invasion), IB, II, or III with serous or clear cell histology
* WHO-performance status 0-2
* WBC ≥ 3.0 x 109/L.
* Platelets ≥ 100 x 109/L.
* Bilirubin ≤ 1.5 x UNL
* ASAT/ALAT ≤ 2.5 x UNL
* Written informed consent

Exclusion criteria:

* Uterine sarcoma (including carcinosarcoma)
* Previous malignancy (except for non-melanomatous skin cancer) < 10 yrs
* Previous pelvic radiotherapy
* Hormonal therapy or chemotherapy for this tumor
* Macroscopic stage II for which Wertheim type hysterectomy (eligible if stage II grade 3 or stage III at pathology)
* Prior diagnosis of Crohn's disease or ulcerative colitis
* Residual macroscopic tumor after surgery
* Creatinine clearance ≤ 60 ml/min (Cockroft) or ≤ 50 ml/min (EDTA clearance, or measured creatinine clearance)
* Impaired cardiac function, prohibiting the infusion of large amounts of fluid during cisplatin therapy
* Peripheral Neuropathy > or = grade 2
* Hearing impairment > or = grade 3, or born deaf

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2006-11-23 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  co-primary endpoint
Failure-free survival | 5 years
  co-primary endpoint

SECONDARY OUTCOMES:
Quality of life by QLQ-C30 v3.0 | 5 years
  Health-related overall quality of life and patient-reported symptom measures
Severe treatment-related morbidity | 5 years
  Acute serious events and SAE and late grade 3-4 complications
Vaginal or pelvic relapse | 5 years
  Both vaginal or pelvic relapse as first failure and total vaginal or pelvic relapse
Distant metastases | 5 years
  Both distant relapse as first failure and total distant relapse

CONTACTS AND LOCATIONS:
Overall Officials: Carien L. Creutzberg, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data will be an option after publication of long-term outcomes and after submission of a research plan with is approved by the with international TMG
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anticipated in 218

REFERENCES:
- [Background] Jameson MG, McNamara J, Bailey M, Metcalfe PE, Holloway LC, Foo K, Do V, Mileshkin L, Creutzberg CL, Khaw P. Results of the Australasian (Trans-Tasman Oncology Group) radiotherapy benchmarking exercise in preparation for participation in the PORTEC-3 trial. J Med Imaging Radiat Oncol. 2016 Aug;60(4):554-9. doi: 10.1111/1754-9485.12447. Epub 2016 Apr 5. PMID 27059658
- [Background] ANZGOG and PORTEC Group; Blinman P, Mileshkin L, Khaw P, Goss G, Johnson C, Capp A, Brooks S, Wain G, Kolodziej I, Veillard AS, O'Connell R, Creutzberg CL, Stockler MR. Patients' and clinicians' preferences for adjuvant chemotherapy in endometrial cancer: an ANZGOG substudy of the PORTEC-3 intergroup randomised trial. Br J Cancer. 2016 Nov 8;115(10):1179-1185. doi: 10.1038/bjc.2016.323. Epub 2016 Oct 20. PMID 27764842
- [Result] de Boer SM, Wortman BG, Bosse T, Powell ME, Singh N, Hollema H, Wilson G, Chowdhury MN, Mileshkin L, Pyman J, Katsaros D, Carinelli S, Fyles A, McLachlin CM, Haie-Meder C, Duvillard P, Nout RA, Verhoeven-Adema KW, Putter H, Creutzberg CL, Smit VTHBM; for PORTEC Study Group. Clinical consequences of upfront pathology review in the randomised PORTEC-3 trial for high-risk endometrial cancer. Ann Oncol. 2018 Feb 1;29(2):424-430. doi: 10.1093/annonc/mdx753. PMID 29190319
- [Result] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Kitchener HC, Nijman HW, Kruitwagen RF, Nout RA, Verhoeven-Adema KW, Smit VT, Putter H, Creutzberg CL; PORTEC study group. Toxicity and quality of life after adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1114-1126. doi: 10.1016/S1470-2045(16)30120-6. Epub 2016 Jul 7. PMID 27397040
- [Result] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Jurgenliemk-Schulz IM, Kitchener HC, Nijman HW, Wilson G, Brooks S, Carinelli S, Provencher D, Hanzen C, Lutgens LCHW, Smit VTHBM, Singh N, Do V, D'Amico R, Nout RA, Feeney A, Verhoeven-Adema KW, Putter H, Creutzberg CL; PORTEC study group. Adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): final results of an international, open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Mar;19(3):295-309. doi: 10.1016/S1470-2045(18)30079-2. Epub 2018 Feb 12. PMID 29449189
- [Result] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, D'Amico R, Fyles A, Baron MH, Jurgenliemk-Schulz IM, Kitchener HC, Nijman HW, Wilson G, Brooks S, Gribaudo S, Provencher D, Hanzen C, Kruitwagen RF, Smit VTHBM, Singh N, Do V, Lissoni A, Nout RA, Feeney A, Verhoeven-Adema KW, Putter H, Creutzberg CL; PORTEC Study Group. Adjuvant chemoradiotherapy versus radiotherapy alone in women with high-risk endometrial cancer (PORTEC-3): patterns of recurrence and post-hoc survival analysis of a randomised phase 3 trial. Lancet Oncol. 2019 Sep;20(9):1273-1285. doi: 10.1016/S1470-2045(19)30395-X. Epub 2019 Jul 22. PMID 31345626
- [Result] Post CCB, de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger NPB, Ledermann JA, Khaw P, D'Amico R, Fyles A, Baron MH, Kitchener HC, Nijman HW, Lutgens LCHW, Brooks S, Jurgenliemk-Schulz IM, Feeney A, Goss G, Fossati R, Ghatage P, Leary A, Do V, Lissoni AA, McCormack M, Nout RA, Verhoeven-Adema KW, Smit VTHBM, Putter H, Creutzberg CL. Long-Term Toxicity and Health-Related Quality of Life After Adjuvant Chemoradiation Therapy or Radiation Therapy Alone for High-Risk Endometrial Cancer in the Randomized PORTEC-3 Trial. Int J Radiat Oncol Biol Phys. 2021 Mar 15;109(4):975-986. doi: 10.1016/j.ijrobp.2020.10.030. Epub 2020 Oct 28. PMID 33129910
- [Result] Leon-Castillo A, de Boer SM, Powell ME, Mileshkin LR, Mackay HJ, Leary A, Nijman HW, Singh N, Pollock PM, Bessette P, Fyles A, Haie-Meder C, Smit VTHBM, Edmondson RJ, Putter H, Kitchener HC, Crosbie EJ, de Bruyn M, Nout RA, Horeweg N, Creutzberg CL, Bosse T; TransPORTEC consortium. Molecular Classification of the PORTEC-3 Trial for High-Risk Endometrial Cancer: Impact on Prognosis and Benefit From Adjuvant Therapy. J Clin Oncol. 2020 Oct 10;38(29):3388-3397. doi: 10.1200/JCO.20.00549. Epub 2020 Aug 4. PMID 32749941
- [Result] Post CCB, Stelloo E, Smit VTHBM, Ruano D, Tops CM, Vermij L, Rutten TA, Jurgenliemk-Schulz IM, Lutgens LCHW, Jobsen JJ, Nout RA, Crosbie EJ, Powell ME, Mileshkin L, Leary A, Bessette P, Putter H, de Boer SM, Horeweg N, Nielsen M, Wezel TV, Bosse T, Creutzberg CL. Prevalence and Prognosis of Lynch Syndrome and Sporadic Mismatch Repair Deficiency in Endometrial Cancer. J Natl Cancer Inst. 2021 Sep 4;113(9):1212-1220. doi: 10.1093/jnci/djab029. PMID 33693762
- [Result] Wortman BG, Post CCB, Powell ME, Khaw P, Fyles A, D'Amico R, Haie-Meder C, Jurgenliemk-Schulz IM, McCormack M, Do V, Katsaros D, Bessette P, Baron MH, Nout RA, Whitmarsh K, Mileshkin L, Lutgens LCHW, Kitchener HC, Brooks S, Nijman HW, Astreinidou E, Putter H, Creutzberg CL, de Boer SM. Radiation Therapy Techniques and Treatment-Related Toxicity in the PORTEC-3 Trial: Comparison of 3-Dimensional Conformal Radiation Therapy Versus Intensity-Modulated Radiation Therapy. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):390-399. doi: 10.1016/j.ijrobp.2021.09.042. Epub 2021 Oct 2. PMID 34610387
- [Result] Khaw P, Do V, Lim K, Cunninghame J, Dixon J, Vassie J, Bailey M, Johnson C, Kahl K, Gordon C, Cook O, Foo K, Fyles A, Powell M, Haie-Meder C, D'Amico R, Bessette P, Mileshkin L, Creutzberg CL, Moore A. Radiotherapy Quality Assurance in the PORTEC-3 (TROG 08.04) Trial. Clin Oncol (R Coll Radiol). 2022 Mar;34(3):198-204. doi: 10.1016/j.clon.2021.11.015. Epub 2021 Dec 11. PMID 34903431
- [Derived] Post CCB, de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Leary A, Ottevanger PB, McCormack M, Khaw P, D'Amico R, Fyles A, Chargari C, Kitchener HC, Do V, Lissoni A, Provencher D, Genestie C, Nijman HW, Whitmarsh K, Jurgenliemk-Schulz IM, Feeney A, Lutgens LCHW, Bouma J, Leon-Castillo A, Nout RA, Putter H, Bosse T, Creutzberg CL. Adjuvant chemoradiotherapy versus radiotherapy alone in women with high-risk endometrial cancer (PORTEC-3): 10-year clinical outcomes and post-hoc analysis by molecular classification from a randomised phase 3 trial. Lancet Oncol. 2025 Oct;26(10):1370-1381. doi: 10.1016/S1470-2045(25)00379-1. Epub 2025 Sep 5. PMID 40921169
- See also: trial website (with protocol and all documents) — http://www.msbi.nl/portec3